## NCT 04247061

## Statistical Analysis Plan

Delivery of a Smoking Cessation Induction Intervention Via Virtual Reality (VR) Headset During a Dental Cleaning: Usability Study There is no plan for formal data analysis, as this is a usability study. We are interested primarily in testing data acquisition procedures, methods, acceptability and satisfaction, and impact on hypothesized theoretical mediators in order to inform and refine the design of a future randomized clinical trial.

We will examine frequency distributions and descriptive statistics of satisfaction data. Questionnaire data will be summarized as means and standard deviations for continuous measures and frequency and proportions for categorical measures. We will compute withingroup mean (or proportion) differences between baseline and the post-video assessment and between baseline and the one-month follow up assessment. Data from text messages will also be summarized as means and standard deviations or frequency and proportions.